CLINICAL TRIAL: NCT00125866
Title: The Effect of Cocoa Polyphenols on Various Cardiovascular Measurements Including Blood Pressure
Brief Title: The Effect of Cocoa Flavonoids on Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: MasterFoods (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NPSW01
Record Dates: First submitted 2005-07-29; First posted 2005-08-02 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2007-04

CONDITIONS: Hypertension
Keywords: randomised double blind trial; blood pressure; cocoa flavonoids
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Behavioral: Flavonoid rich or flavonoid depleted chocolate drink

SUMMARY:
The purpose of this study is to compare the effects on blood pressure of a daily intake of a flavonoid-rich cocoa drink with that of the same drink from which the flavonoids have been largely extracted.

DETAILED DESCRIPTION:
Flavonoids are natural substances found in fruits and vegetables, tea and red wine. The investigators know that people who eat a diet rich in these foods are less likely to have heart disease. This, in part, may be due to the blood pressure lowering effect of flavonoids. Cocoa beans are a rich natural source of flavonoids. Unfortunately when cocoa is made into chocolate most of the flavonoids are destroyed. The aim of this study is to find out the effect of cocoa flavonoids on blood pressure after 12 weeks of daily consumption of a specially prepared chocolate drink that is rich in flavonoids.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of any age.
* Diagnosis of hypertension and on antihypertensive treatment.
* Stable blood pressure that has reached the British Hypertension Society (BHS) audit standard (<150/90mmHg).

Exclusion Criteria:

* Participation in another clinical trial.
* Any reason to suspect that the patient will not comply with drinking a chocolate beverage every day for the trial duration.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2005-09; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Difference in mean 24 hour ambulatory blood pressure

SECONDARY OUTCOMES:
Difference in cholesterol
Difference in glucose
Difference in insulin
Difference in echocardiogram
Difference in pulse wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: Neil R Poulter, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, Paddington, London, United Kingdom